CLINICAL TRIAL: NCT00205504
Title: Oral Contraceptives in the Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM4060
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2012-05-07 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Metabolic Syndrome X; Insulin Resistance; Obesity; Cardiovascular Diseases
Keywords: Inflammatory markers, oral contraceptions, obesity, metabolic syndrome X
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Obesity; Cardiovascular Diseases | interventions — Moxifloxacin

ARMS (3):
- Obese women with metabolic syndrome (Active Comparator)
  Interventions: Drug: Ortho Tri Cyclen
- Obese women without metabolic syndrome (Active Comparator)
  Interventions: Drug: Ortho Tri Cyclen
- lean women without metabolic syndrome (Active Comparator)
  Interventions: Drug: Ortho Tri Cyclen

INTERVENTIONS:
Drug: Ortho Tri Cyclen — Ortho Tri Cyclen, one tablet daily, for 6 cycles

SUMMARY:
Oral contraceptives (OCs) are the most widely used method of reversible birth control. However, the long-term cardiovascular safety of the widely used low-dose OCs (ethinyl-estradiol < 50 mcg) is still debated. Although cardiovascular events are rare in young women whether they use OCs or not, the risks of myocardial infarction and ischemic stroke are increased among users of OCs who have conventional cardiovascular risk factors such as use of tobacco, diabetes or hypercholesterolemia. However, the risk of cardiovascular events in OC users with emerging cardiovascular risk factors (such as obesity and the metabolic syndrome) have not been investigated. Recently, the metabolic syndrome has been linked with the risk of cardiovascular disease. The syndrome is a clustering of risk factors in a single individual, and its underlying cause may be insulin resistance. Whether the metabolic syndrome predicts a higher cardiovascular risk in OC users has not been studied. This is a critical problem because the metabolic syndrome is prevalent in 24% of adults. Until the cardiovascular risks in users of OC are clearly defined, the appropriate use of OC with the least harm would not be possible.

The investigator's long-term goal is to understand the best way to prevent and treat cardiovascular disease in women. The objective of this particular project is to obtain pilot data on the extent to which the metabolic syndrome and obesity affects glucose metabolism and cardiovascular risks in women taking OCs. The researchers hypothesize that women with metabolic syndrome and obese women will have worsened glucose metabolism and elevated cardiovascular risks associated with OC use, when compared to normal weight women without the metabolic syndrome. Results of this study will clarify the risk factors for cardiovascular events in women taking OCs, and will serve as pilot data for a National Institutes of Health (NIH) proposal. Once the cardiovascular risk factors of OC users are understood, clinicians can make better informed decisions about contraceptive choices for their patients.

ELIGIBILITY:
Inclusion Criteria:

1. Acceptable health based on interview, medical history, physical examination, and laboratory tests (comprehensive metabolic panel - SMA20, and complete blood count - CBC);
2. Have not taken oral contraceptives (OCs) in the past 3 months;
3. Ability to comply with the requirements of the study;
4. Ability and willingness to provide signed, witnessed informed consent. In addition, women with the metabolic syndrome must meet the National Cholesterol Education Program (NCEP) defined criteria of the metabolic syndrome, that is, having at least 3 of the 5 factors:

   1. increased waist circumference > 35 inches,
   2. hypertriglyceridemia ≥ 150 mg/dL,
   3. low high-density lipoprotein (HDL) cholesterol < 50 mg/dL in women,
   4. hypertension (≥ 130/≥ 85 mmHg),
   5. fasting glucose ≥ 100 mg/dL.

Obese women with or without the metabolic syndrome should have a Body Mass Index (BMI) > 30 kg/m2 and lean women should have a Body Mass Index BMI < 25 kg/m2.

Exclusion Criteria:

1. Diabetes mellitus by fasting glucose or a 2-hour oral glucose tolerance test (OGTT);
2. Clinically significant pulmonary, cardiac (including but not limited to ischemic heart disease, stable/unstable angina, and congestive heart failure), renal, hepatic, cholestatic, neurologic, psychiatric, infectious, and malignant disease (other than melanoma skin cancer);
3. History of thromboembolism, myocardial infarction, cerebrovascular accident, vascular disease, known coagulopathy, prolonged immobilization, or recent major surgery (within past 6 months);
4. Systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 100 mmHg (mild hypertension is not an exclusion criterion);
5. History of breast cancer, migraine headaches, or age ≥ 35 years and smoker of ≥ 20 cigarettes/day;
6. Use of metformin, thiazolidinediones, anti-hyperlipidemic drugs, anti-hypertensive drugs, glucocorticoids, or anti-androgens (spironolactone, flutamide, etc.) within 3 months;
7. Documented or suspected illicit drug abuse or alcoholism within one year;
8. Ingestion of any investigational drugs within 3 months prior to the study onset; and
9. Pregnancy or lactation (≤ 6 weeks postpartum);
10. Hematocrit < 33g/dL. These exclusion criteria are based on study requirements and also go beyond guidelines for OC use published by the World Health Organization.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2005-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kai I Cheang, Pharm.D., Principal Investigator — Virginia Commonwealth University; John E Nestler, M.D., Study Director — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University General Clinical Research Center, Richmond, Virginia, United States

REFERENCES:
- [Result] Cheang KI, Essah PA, Sharma S, Wickham EP 3rd, Nestler JE. Divergent effects of a combined hormonal oral contraceptive on insulin sensitivity in lean versus obese women. Fertil Steril. 2011 Aug;96(2):353-359.e1. doi: 10.1016/j.fertnstert.2011.05.039. Epub 2011 Jun 15. PMID 21676394

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 46 completed informed consent, only 36 initiated the study. Among The participants who did not begin the study were lost to follow-up prior to beginning the protocol, were no shows, or withdrew from the study before beginning study procedures.
Groups:
- Obese Women: Women with Body Mass Index (BMI) >30 kg/m².
  Note: Only two arms were analyzed for the results. Women who were candidates for taking oral contraceptive pills and had the metabolic syndrome could not be recruited. That is because some inclusion criteria for metabolic syndrome are actually exclusion criteria for safe oral contraceptive use.
- Lean Women: Women with Body Mass Index)BMI <25 kg/m²
Period: Overall Study
Arm/Group | Obese Women | Lean Women
Started | 21 | 15
Completed | 14 | 15
Not Completed | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obese Women | Lean Women | Total
Number analyzed (Participants) | 21 | 15 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 15 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (6.9) | 21.4 (2.3) | 23.4 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 36
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 15 | 36

OUTCOME MEASURES:

1. Primary Outcome: Changes in Insulin Sensitivity Associated With Oral Contraceptive (OC) Use Compared Among (1) Obese Women and (2) Lean Women
Description: Insulin sensitivity was assessed by frequent sampling intravenous glucose tolerance test (FSIVGTT).
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mIU/L
Groups:
- Obese Women: Women with Body Mass Index (BMI) >30 kg/m²
- Lean Women: Women with Body Mass Index (BMI) <25 kg/m²
Arm/Group | Obese Women | Lean Women
Number analyzed (Participants) | 14 | 15
mIU/L
  Baseline Insulin sensitivity | 4.36 (2.32) | 6.62 (3.69)
  6 months Insulin sensitivity | 3.82 (3.12) | 8.23 (3.30)

2. Secondary Outcome: Changes in Lipid Profile Compared Associated With OC Use Among (1) Obese Women and (2) Lean Women
Description: The lipid profile is assessed through blood sample analysis for low-density lipoprotein (LDL), Triglycerides and high-density lipoprotein (HDL).
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Obese Women | Lean Women
Number analyzed (Participants) | 14 | 15
mg/dL
  Baseline LDL | 95 (18.4) | 84 (24.3)
  6 months LDL | 113 (25.2) | 104 (26.1)
  Baseline Triglycerides | 72 (50.3) | 72 (52.0)
  6 months Triglycerides | 83 (51.1) | 106 (52.9)
  Baseline HDL | 51 (10.7) | 53 (10.0)
  6 months HDL | 58 (12.4) | 61 (12.8)

3. Secondary Outcome: Inflammatory Marker Changes, High Sensitive C-reactive Protein (Hs-CRP) and Adiponectin, Associated With OC Use Compared Among (1) Obese Women and (2) Lean Women
Description: Inflammatory markers are assessed through blood analysis for C-reactive protein (hs-CRP) and adiponectin.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Obese Women | Lean Women
Number analyzed (Participants) | 14 | 15
ng/mL
  Baseline Hs-CRP | 4908.76 (5215.07) | 2050.77 (4748.75)
  6 months Hs-CRP | 6207.76 (4566.8) | 2266.02 (3443.3)
  Baseline Adiponectin | 17568.86 (5680.86) | 21976.53 (8322.05)
  6 months Adiponectin | 18408.43 (4934.39) | 22221.36 (11160.97)

4. Secondary Outcome: Changes in Estrogen Metabolites (Plasma) Associated With OC Use Compared Among (1) Obese Women and (2) Lean Women
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Obese Women | Lean Women
Number analyzed (Participants) | 14 | 15
pg/mL
  Baseline 16aE1 | 314.76 (179.73) | 317.47 (159.8)
  6 months 16aE1 | 421.6 (286.57) | 383.39 (452.98)
  Baseline 2ME1 | 25.92 (11.03) | 32.39 (9.3)
  6 months 2ME1 | 52.84 (54.29) | 45.58 (23.83)
  Baseline 4ME1 | 5.26 (3.58) | 4.45 (3.13)
  6 months 4ME1 | 6.1 (3.29) | 7.42 (8.55)
  Baseline 2ME2 | 1.48 (1.06) | 0.91 (0.82)
  6 months 2ME2 | 1.5 (1.11) | 1.74 (2.15)
  Baseline E1 | 217.23 (170.88) | 245.99 (128.41)
  6 months E1 | 315.03 (339.15) | 227.4 (271.6)
  Baseline 4ME2 | 0.73 (0.55) | 0.59 (0.54)
  6 months 4ME2 | 0.89 (0.79) | 1.14 (1.41)
  Baseline E2 | 34.11 (15.61) | 36.796 (17.28)
  6 months E2 | 74.73 (117.52) | 47.32 (61.82)
  Baseline 2OHE1 | 101.07 (126.04) | 85.62 (48.08)
  6 months 2OHE1 | 135.95 (220.24) | 57.96 (70.02)
  Baseline 2OHE2 | 9.81 (5.85) | 8.01 (3.62)
  6 months 2OHE2 | 11.55 (21.74) | 6.05 (4.69)
  Baseline 4OHE1 | 33.78 (16.52) | 33.98 (25.86)
  6 months 4OHE1 | 27.29 (25.65) | 29.12 (15.08)
  Baseline Total plasma | 1068 (472.78) | 1022.16 (295.61)
  6 months Total plasma | 1342.21 (1166.36) | 1007.89 (977.81)

5. Secondary Outcome: Changes in Waist-to-Hip Ratio Associated With OC Use Compared Among (1) Obese Women and (2) Lean Women
Description: Waist-to-hip ratio is assessed through calculated ratio of waist and hip circumference.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Obese Women | Lean Women
Number analyzed (Participants) | 14 | 15
ratio
  Baseline Waist-Hip Ratio | 0.79 (0.059) | 0.73 (0.027)
  6 months Waist-Hip Ratio | 0.81 (0.057) | 0.73 (0.057)

6. Secondary Outcome: Inflammatory Marker Changes (MCP-1) Associated With OC Use Compared Among (1) Obese Women and (2) Lean Women
Description: Inflammatory marker is assessed through blood analysis for Monocyte chemotactic protein-1 (MCP-1).
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Obese Women: Women with BMI >30 kg/m²
- Lean Women: Women with BMI >25 kg/m²
Arm/Group | Obese Women | Lean Women
Number analyzed (Participants) | 14 | 15
pg/mL
  Baseline MCP-1 | 209.56 (125.92) | 156.14 (36.29)
  6 months MCP-1 | 219.86 (159.85) | 206.66 (76.15)

7. Secondary Outcome: Changes in Blood Pressure Associated With OC Use Compared Among (1) Obese Women and (2) Lean Women
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Obese Women | Lean Women
Number analyzed (Participants) | 14 | 15
mm Hg
  Baseline Systolic Blood Pressure | 121.1 (3.2) | 105.7 (8.6)
  6 months Systolic Blood Pressure | 123.5 (11.7) | 106.5 (12.2)
  Baseline Diastolic Blood Pressure | 74.4 (1.8) | 68.0 (3.7)
  6 months Diastolic Blood Pressure | 73.4 (6.6) | 66.5 (6.8)

8. Secondary Outcome: Changes in Body Mass Index (BMI) Associated With OC Use Compared Among (1) Obese Women and (2) Lean Women
Description: Body Mass Index is a calculation of height and weight: kg/m²
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: kg/m²
Arm/Group | Obese Women | Lean Women
Number analyzed (Participants) | 14 | 15
kg/m²
  Baseline BMI | 37.1 (6.7) | 21.3 (1.8)
  6 months BMI | 37.6 (4.7) | 21.4 (4.9)

9. Secondary Outcome: Changes in Waist Circumference Associated With OC Use Compared Among (1) Obese Women and (2) Lean Women
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Obese Women | Lean Women
Number analyzed (Participants) | 14 | 15
cm
  Baseline Waist circumference | 100.0 (14.4) | 70.2 (4.1)
  6 months Waist circumference | 101.0 (10.5) | 70.9 (10.7)

10. Secondary Outcome: Inflammatory Marker Changes, Soluble Vascular Cell Adhesion Molecule (sVCAM) and Soluble Intercellular Adhesion Molecule (sICAM), Associated With OC Use Compared Among (1) Obese Women and (2) Lean Women
Description: These inflammatory markers are assessed through blood analysis of Soluble Vascular Cell Adhesion Molecule (sVCAM) and soluble intercellular adhesion molecule (sICAM).
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Obese Women | Lean Women
Number analyzed (Participants) | 14 | 15
ng/mL
  Baseline sVCAM | 905 (190.63) | 1139.6 (159.57)
  6 months sVCAM | 880.14 (180.08) | 1003.29 (256.62)
  Baseline sICAM | 163.34 (50.44) | 182.11 (91.17)
  6 months sICAM | 163.2 (27.71) | 160.21 (74.88)

ADVERSE EVENTS:
Arm/Group | Obese Women | Lean Women
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/15
Other Adverse Events (participants affected / at risk) | 2/21 | 2/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Obese Women (N=21) | Lean Women (N=15)
Gallstones removal (Gastrointestinal disorders) | 1 | 0 — Subject had gallstones removed during study, and continued study.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Obese Women (N=21) | Lean Women (N=15)
Tiredness (Injury, poisoning and procedural complications) | 0 | 1 — Subject felt tired during her last day of study and did not desire to continue that morning's study procedure.
Pain with venipuncture (Injury, poisoning and procedural complications) | 0 | 1 — Subject withdrew withdrew after the first two mornings of study because of pain associated with venipuncture.
Phlebitis due to catheter insertion (Injury, poisoning and procedural complications) | 1 | 0 — Subject experienced phlebitis at the site of catheter insertion. Subject was discontinued from the study by investigator.
Dizziness due to Ortho Tricyclen (Injury, poisoning and procedural complications) | 1 | 0 — Subject withdrew after 1 day of study medication (Ortho Tricyclen)due to dizziness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes